CLINICAL TRIAL: NCT05851482
Title: NOVEL HIGH-RESOLUTION MANOMETRY SCORE FOR THE DIAGNOSIS OF GASTRO-ESOPHAGEAL REFLUX DISEASE
Brief Title: Validation of HRM Score for the GERD Diagnosis
Acronym: HRM nomogram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: University of Milan (Other); Medical University of Vienna (Other); Washington University School of Medicine (Other); University of Pisa (Other); Swedish Medical Center (Other); Hospital Universiti Sains Malaysia (Other); University of Campania Luigi Vanvitelli (Other); Universita degli Studi di Genova (Other); Jikei University School of Medicine (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); University of Athens (Other)
Responsible Party: Principal Investigator, Stefano Siboni, Medical Doctor, IRCCS Policlinico S. Donato
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HRM Nomogram GERD
Record Dates: First submitted 2023-04-29; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Gastro Esophageal Reflux
Keywords: High Resolution Manometry; Gastroesophageal reflux disease; Esophagogastric junction; Inta-abdominal pressure; Straight leg raise maneuver
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Prospective descriptive study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GERD (Experimental): Patients with GERD symptoms
  Interventions: Diagnostic Test: High resolution manometry

INTERVENTIONS:
Diagnostic Test: High resolution manometry — Standard chicago classification 4.0 HRM protocol

SUMMARY:
The goal of this prospective study is to validate a high resolution manometry score to predict pathologic GERD in patients with reflux symptoms. The main question it aims to answer is:

Is it possible to predict GERD on high resolution manometry? Participants will be asked to undergo high resolution manometry and pH-study

DETAILED DESCRIPTION:
According to recent guidelines, high resolution manometry (HRM) has an ancillary role in the diagnosis of gastro-esophageal reflux disease (GERD). A recent multicenter study demonstrated the effectiveness of the straight leg raise (SLR) maneuver in predicting GERD, thus increasing the diagnostic value of HRM in patients with suspected pathological reflux. HRM parameters associated with GERD include esophageal body hypomotility such as ineffective esophageal motility (IEM), and esophagogastric junction (EGJ) metrics, particularly the EGJ contractile integral (EGJ-CI) that takes into consideration the presence or absence of a hiatal hernia (HH), and a hypotensive lower esophageal sphincter (LES). The combination of these four parameters might help to predict or exclude true GERD in patients undergoing HRM with the suspicion of GERD.

In this multicenter international prospective study, we aimed to build a score to predict pathological esophageal acid exposure time (AET>6%).

ELIGIBILITY:
Inclusion Criteria:

* HRM and wireless pH-study or catheter pH-impedance study performed for persistent GERD symptoms off proton-pump inhibitor (PPI) within two weeks of each other,
* SLR maneuver performed at the end of HRM

Exclusion Criteria:

* Body mass index (BMI) >35 Kg/m2
* prior esophageal surgery
* paraesophageal hiatal hernia
* eosinophilic esophagitis
* scleroderma
* esophageal achalasia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-29 (Actual)

PRIMARY OUTCOMES:
HRM score | From date of inclusion in the study until the diagnosis of GERD, up to 2 months
  HRM score is based on EJG type, ineffective esophageal motility, straight leg raise maneuver and EGJ contractile integral

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Siboni, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siboni S, Kristo I, Rogers BD, De Bortoli N, Hobson A, Louie B, Lee YY, Tee V, Tolone S, Marabotto E, Visaggi P, Haworth J, Ivy M, Greenan G, Facchini C, Masuda T, Yano F, Perry K, Balasubramanian G, Theodorou D, Triantafyllou T, Cusmai L, Boveri S, Schoppmann SF, Gyawali CP, Bonavina L. Improving the Diagnostic Yield of High-Resolution Esophageal Manometry for GERD: The "Straight Leg-Raise" International Study. Clin Gastroenterol Hepatol. 2023 Jul;21(7):1761-1770.e1. doi: 10.1016/j.cgh.2022.10.008. Epub 2022 Oct 19. PMID 36270615
- [Derived] Siboni S, Sozzi M, Kristo I, Boveri S, Rogers BD, De Bortoli N, Hobson A, Louie BE, Lee YY, Tolone S, Marabotto E, Visaggi P, Haworth J, Ivy ML, Greenan G, Masuda T, Penagini R, Barcella B, Coletta M, Theodorou D, Triantafyllou T, Facchini C, Tee V, Bonavina L, Cusmai L, Schoppmann SF, Savarino E, Asti E, Gyawali CP. The Milan score: A novel manometric tool for a more efficient diagnosis of gastro-esophageal reflux disease. United European Gastroenterol J. 2024 Jun;12(5):552-561. doi: 10.1002/ueg2.12565. Epub 2024 Mar 27. PMID 38536701